CLINICAL TRIAL: NCT07154069
Title: Adaptive Immunotherapy for Locoregional Nasopharyngeal Carcinoma: a Randomized, Controlled, Multicenter, Phase 3 Clinical Trial
Brief Title: Adaptive Immunotherapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ling-Long Tang, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-489-01
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
MeSH Terms: interventions — Capecitabine; Chemoradiotherapy; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low risk arm 1 (Experimental): Radiotherapy alone
  Interventions: Radiation: Radical radiotherapy of nasopharynx and neck; Drug: Toripalimab
- Low risk arm 2 (Active Comparator): Concurrent chemoradiotherapy
  Interventions: Radiation: Radical radiotherapy of nasopharynx and neck; Drug: Concurrent chemoradiotherapy (cCRT); Drug: Toripalimab
- High risk arm 1 (Experimental): Adjuvant capecitabine and immunotherapy after concurrent chemoradiotherapy
  Interventions: Radiation: Radical radiotherapy of nasopharynx and neck; Drug: Capecitabine; Drug: Concurrent chemoradiotherapy (cCRT); Drug: Toripalimab
- High risk arm 2 (Active Comparator): Adjuvant immunotherapy after concurrent chemoradiotherapy
  Interventions: Radiation: Radical radiotherapy of nasopharynx and neck; Drug: Concurrent chemoradiotherapy (cCRT); Drug: Toripalimab

INTERVENTIONS:
Radiation: Radical radiotherapy of nasopharynx and neck — Radical radiotherapy of nasopharynx and neck
Drug: Capecitabine — Adjuvant metronomic capecitabine (650 mg/m² twice daily) for one year
  Arms: High risk arm 1
Drug: Concurrent chemoradiotherapy (cCRT) — Concurrent chemoradiotherapy
  Arms: High risk arm 1; High risk arm 2; Low risk arm 2
Drug: Toripalimab — Adjuvant Toripalimab (240mg day1, Q3W )

SUMMARY:
1. To assess whether radiotherapy alone is non-inferior to concurrent chemoradiotherapy with respect to event-free survival and superior in reducing treatment-related nausea in low-risk locoregionally advanced nasopharyngeal carcinoma patients who achieve complete or partial response and undetectable serum EBV-DNA following induction chemoimmunotherapy.
2. To evaluate whether adjuvant capecitabine and immunotherapy after concurrent chemoradiotherapy improves event-free survival compared to adjuvant immunotherapy in high-risk locoregionally advanced nasopharyngeal carcinoma patients with stable disease or detectable serum EBV-DNA after induction chemoimmunotherapy.

DETAILED DESCRIPTION:
Recent trials have demonstrated that for patients with locoregionally advanced nasopharyngeal carcinoma (NPC), the addition of immnotherapy to standard induction chemotherapy followed by concurrent chemoradiotherapy significantly improves event-free survival (EFS) (NCT03700476 and NCT03427827). However, current trials on immnotherapies lack specific biomarkers for risk stratification and adaptive treatment strategies.

Epstein-Barr virus (EBV) is closely associated with the development of NPC. Cell-free EBV-DNA released by NPC cells can be detected in peripheral blood and has been strongly correlated with patient prognosis. Prospective clinical trials (NCT03855020 and NCT04907370) have confirmed that patients with undetectable EBV-DNA after induction therapy exhibit significantly better EFS compared to those with detectable post-induction EBV-DNA.

Among low-risk patients with undetectable EBV-DNA after induction therapy, the 3-year EFS rate exceeds 90%. However, the combination of immunotherapy with concurrent cisplatin-based chemoradiotherapy also leads to significant treatment-related toxicities, with 74% of patients experiencing grade 3 or higher adverse events. Therefore, there is an urgent need to explore novel treatment strategies aimed at reducing toxicity in this patient population. Recent phase 3 multicenter randomized trials have demonstrated that de-intensification strategies omitting concurrent cisplatin chemotherapy significantly reduce treatment-related toxicities in both early-stage (NCT02633202) and locoregionally advanced NPC (NCT04907370), with reductions in grade 3 or higher adverse events by 29% and 11%, respectively.

Among high-risk patients with positive EBV-DNA after induction therapy, even with the combination of immuotherapy, the 3-year EFS remains suboptimal, ranging from 65% to 80%. There is a critical need for treatment intensification strategies to improve outcomes in this group. A recently completed multicenter, randomized, phase 3 trial (NCT02958111) demonstrated that adjuvant metronomic capecitabine (650 mg/m² twice daily) for one year following standard induction chemotherapy and concurrent chemoradiotherapy significantly improved 3-year EFS from 75.7% to 85.3% in high-risk locoregionally advanced NPC patients, with a manageable toxicity profile.

Therefore, the investigators propose the following scientific hypothesis: in low-risk patients who achieve complete or partial response and undetectable serum EBV-DNA following induction chemoimmunotherapy, radiotherapy alone can reduce the incidence of treatment-related adverse effects, without reducing survival; in high-risk patients with stable disease or detectable serum EBV-DNA, adjuvant capecitabine and immunotherapy can improve survival.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years;
* Newly diagnosed, pathologically confirmed non-keratinizing carcinoma (according to WHO criteria);
* Locoregionally advanced nasopharyngeal carcinoma (Stage II-III) as defined by the 9th edition of the American Joint Committee on Cancer (AJCC) staging system;
* ECOG performance status: 0-1;
* Adequate bone marrow function: white blood cell count > 4 × 10⁹/L, hemoglobin > 90 g/L, platelet count > 100 × 10⁹/L;
* Normal renal and hepatic function: total bilirubin ≤ 1.5 × upper limit of normal (ULN); aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; creatinine clearance ≥ 60 mL/min;
* Normal thyroid function, amylase, lipase, pituitary function;
* Completion of 3 cycles of GP regimen induction chemotherapy combined with PD-1 inhibitor immunotherapy;
* Patients must provide signed informed consent and be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures;
* Female participants of childbearing potential must agree to use reliable contraceptive methods (e.g., condoms, regular use of oral contraceptives as prescribed) from screening until one year after treatment.

Exclusion Criteria:

* T3N0-1, according to the American Joint Committee on Cancer (AJCC) Staging System, 9th Edition;
* Disease progression after induction therapy;
* Hepatitis B surface antigen (HBsAg) positive with HBV DNA >1×10³ copies/mL, or anti-hepatitis C virus (HCV) antibody positive;
* Anti-HIV antibody positive or diagnosed with acquired immunodeficiency syndrome (AIDS);
* Active tuberculosis;
* Active, known, or suspected autoimmune disease. Exceptions include type 1 diabetes, hypothyroidism requiring hormone replacement therapy, and skin disorders not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia);
* History of interstitial lung disease or pneumonia requiring oral or intravenous steroid treatment within the past year;
* Chronic systemic glucocorticoid therapy or any other form of immunosuppressive therapy. Subjects using inhaled or topical corticosteroids are eligible;
* Uncontrolled cardiac disease;
* Pregnant or lactating women;
* History or current diagnosis of another malignancy, except for adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, or papillary thyroid carcinoma;
* Known allergy to macromolecular protein preparations or any component of toripalimab;
* Active infection requiring systemic treatment within one week prior to enrollment;
* Administration of a live vaccine within 30 days before the first dose of toripalimab;
* History of organ transplantation;
* Contraindications to MRI examination, which would prevent the completion of required imaging;
* Any other condition deemed by the investigators to potentially compromise patient safety or compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 year
  The primary endpoint was event-free survival from randomisation to disease recurrence (locoregional or distant) or death from any cause in the intention-to-treat population.
Incidence rates of vomiting as assessed by CTCAE v5.0 | 3 year
  In the low-risk arm, the primary outcome included the incidence rates of vomiting (evaluated according to the Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).

SECONDARY OUTCOMES:
Overall survival | 3 year
  The secondary endpoint include overall survivall from randomisation to death from any cause in the intention-to-treat population.
Locoregional relapse-free survival | 3 year
  The secondary endpoint include locoregional relapse-free survival from randomisation to local and/or regional relapse or death from any cause in the intention-to-treat population.
Distant metastasis-free survival | 3 year
  The secondary endpoint include distant metastasis-free survival from randomisation to distant metastasis or death from any cause in the intention-to-treat population.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 year
  Acute and late treatment-related adverse events will be assessed by the CTCAE v 5.0(Common Terminology Criteria for Adverse Events, version 5.0).
Number of participants with treatment-related adverse events as assessed by RTOG/EORTC System | 3 year
  Acute and late treatment-related adverse events will be documented according to RTOG/EORTC System.
Patient's quality-of-life as assessed by EORTC QLQ-C30 | 3 year
  The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) version 3.0 questionnaires will be used to assess quality-of-life
Patient's quality-of-life as assessed by QLQ-H&N35 v1.0 | 3 year
  Using Quality-of-Life Head and Neck 35 items (QLQ-H&N35) version 1.0 questionnaires
Patient-reported tolerability as assessed by PRO-CTCAE v1.0 | 3 year
  Tolerability was assessed from patients' subjective experience using PRO-CTCAE (version 1.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No